CLINICAL TRIAL: NCT03259542
Title: A Phase 1, Open-Label, Drug-Drug Interaction Study in Healthy Subjects to Determine the Effects of a Strong Inhibitor (Itraconazole) of Cytochrome P450 3A on Exposure to Mifepristone and Its Metabolites
Brief Title: Mifepristone Drug-Drug Interaction Study With CYP3A Inhibitor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C1073-38
Record Dates: First submitted 2017-08-07; First posted 2017-08-23 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2017-10

CONDITIONS: Drug Interaction Potentiation; Healthy
MeSH Terms: interventions — Mifepristone; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Mifepristone 300 MG alone or Mifepristone 300 MG with Itraconazole 100 MG will be administered.
  Interventions: Drug: Mifepristone 300 MG; Drug: Itraconazole 100 MG

INTERVENTIONS:
Drug: Mifepristone 300 MG — mifepristone 300 MG (4 tablets) orally for a total of 1200 mg a day for 14 days; then mifepristone 300 mg (3 tablets) orally for a total of 900 mg a day for 28 days
Drug: Itraconazole 100 MG — itraconazole 100 MG (2 capsules) orally for a total of 200 MG for the last 14 days of mifepristone dosing

SUMMARY:
This is a Phase 1, single-center, fixed-sequence, open label, drug-drug interaction study of the effect of multiple daily doses of oral itraconazole 200 mg, a strong inhibitor of CYP3A, given with mifepristone 900 mg QD, in healthy male subjects, where all drug administrations are given after a meal.

ELIGIBILITY:
Inclusion Criteria:

* Be healthy
* Have a BMI of 18 to 32 kg/m2, inclusive and body weight more than 50 kg (110 pounds)
* Be judged to be in good health, based on the results of medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory findings
* Have suitable veins for multiple venipuncture/cannulation

Exclusion Criteria:

* Have multiple drug allergies, or be allergic to any of the components of mifepristone or itraconazole
* Have a condition that could be aggravated by glucocorticoid blockade (eg, asthma, any chronic inflammatory condition)
* In the 1 year before study drug administration, have a history of drug or alcohol abuse
* In the 6 calendar months before study drug administration, on average

  * Have smoked more than 5 cigarettes/day
  * Have consumed more than 21 units of alcohol/week (1 unit/drink = 5 ounces of wine, or 12 ounces of beer, or 1.5 ounces of hard liquor)
* In 2 months prior to study drug administration, have donated/lost blood or plasma in excess of 400 mL
* In the 30 days before study drug administration, have participated in another clinical trial of a new chemical entity or a prescription medicine

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Not based on self-representation of gender identity
Enrollment: 33 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Cmax of mifepristone at Day 42 compared to Day 28 | Day 42 compared to Day 28
  Maximum (peak) plasma drug concentration (Cmax)
AUC0-24 of mifepristone at Day 42 compared to Day 28 | Day 42 compared to Day 28
  Area under the plasma concentration-time curve from zero to 24 hours (AUC0-24)

SECONDARY OUTCOMES:
Cmax of mifepristone at Day 42 compared to Day 14 | Day 42 compared to Day 14
AUC0-24 of mifepristone compared to Day 14 | Day 42 compared to Day 14
T1/2 of mifepristone | Days 14 and 28
  Elimination half-life (T1/2)
Ctrough of mifepristone | Days 1 through 28
  Trough plasma concentration (measured concentration at the end of a dosing interval at steady state [taken directly before next administration]) (Ctrough)

CONTACTS AND LOCATIONS:
Overall Officials: Ada Lee, MD, Study Director — Corcept Therapeutics
Locations (1):
- SeaView Research, Miami, Florida, United States